CLINICAL TRIAL: NCT06963736
Title: WatchWell: Simple and Practical Strategies to Reduce the Negative Health Impact of Sedentary Screen Time
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Matthew P Buman, PhD, Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00021203
Record Dates: First submitted 2025-04-29; First posted 2025-05-09 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Sedentary Time; Cardiovascular Diseases; Prediabetes; Obesity
Keywords: sedentary screen time; blue light; sedentary behavior; standing; crossover design; glucose metabolism
MeSH Terms: conditions — Sedentary Behavior; Cardiovascular Diseases; Prediabetic State; Obesity | interventions — Blue Light; Eating; Standing Position

STUDY DESIGN:
Intervention Model Description: This is a crossover trial where study participants will experience two conditions following a baseline usual behavior condition. All study participants will experience two of three following conditions: avoiding dietary intake after 8p; blocking blue-light exposure after 8p; and breaking up prolonged sitting with standing after 5p.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Blue light-Eating (Experimental): Intervention 1: Participants will be encouraged to wear blue light blocking glasses at 8pm until bed time.
  Intervention 2: Participants will be encouraged to stop eating at 8pm.
  Interventions: Behavioral: Blue light; Behavioral: Eating
- Blue light-standing (Experimental): Intervention 1: Participants will be encouraged to wear blue light blocking glasses at 8pm until bed time.
  Intervention 2: Participants will be sent notifications each hour on the hour from 5pm until bed time to stand for 10 minutes that hour.
  Interventions: Behavioral: Blue light; Behavioral: Standing
- Eating-Standing (Experimental): Intervention 1: Participants will be encouraged to stop eating at 8pm. Intervention 2: Participants will be sent notifications each hour on the hour from 5pm until bed time to stand for 10 minutes that hour.
  Interventions: Behavioral: Eating; Behavioral: Standing
- Eating-Blue Light (Experimental): Intervention 1: Participants will be encouraged to stop eating at 8pm. Intervention 2: Participants will be encouraged to wear blue light blocking glasses at 8pm until bed time.
  Interventions: Behavioral: Blue light; Behavioral: Eating
- Standing-Blue Light (Experimental): Intervention 1: Participants will be sent notifications each hour on the hour from 5pm until bed time to stand for 10 minutes that hour.
  Intervention 2: Participants will be encouraged to wear blue light blocking glasses at 8pm until bed time.
  Interventions: Behavioral: Blue light; Behavioral: Standing
- Standing-Eating (Experimental): Intervention 1: Participants will be sent notifications each hour on the hour from 5pm until bed time to stand for 10 minutes that hour.
  Intervention 2: Participants will be encouraged to stop eating at 8pm.
  Interventions: Behavioral: Eating; Behavioral: Standing

INTERVENTIONS:
Behavioral: Blue light — Blue light blocking glasses use and discouraged late night eating.
  Arms: Blue light-Eating; Blue light-standing; Eating-Blue Light; Standing-Blue Light
Behavioral: Eating — Encouraged not to eat past 8pm.
  Arms: Blue light-Eating; Eating-Blue Light; Eating-Standing; Standing-Eating
Behavioral: Standing — Encouraged to stand for 10 minutes per hour each out from 5pm to bed time.
  Arms: Blue light-standing; Eating-Standing; Standing-Blue Light; Standing-Eating

SUMMARY:
The purpose of this study is to determine the feasibility, acceptability, efficacy, and participant adherence in using home-based technologies and wearable devices and simple, practical strategies to reduce the negative impact that evening screen time may have on your health.

DETAILED DESCRIPTION:
Sedentary screen time (SST) is the most common discretionary activity among all US age and race/ethnic groups. SST is associated with poor health outcomes, including cardiovascular disease (CVD). Recreational SST (rSST) is 2-3X more detrimental to health than other forms of sedentary behavior (e.g., workplace sitting, traveling). Elucidating the mechanisms that lead to elevated harm resulting from rSST is critical. Impact of the COVID-19 pandemic to increase rSST amplifies the urgency of understanding rSST-related mechanisms that lead to detrimental health outcomes. Previous SST studies are limited in scope of intervention and outcomes. There are vital gaps in knowledge about how rSST and rSST-associated behaviors lead to increased CVD risk. Interventions applied in ecologically valid, real-world settings are urgently needed to develop the most potent interventions that address and attenuate critical mechanistic pathways that mediate rSST-associated health risks. WatchWell is a pilot study designed to achieve three important goals that will support our obtaining funding for this research and is responsive to reviewer comments on our previously submitted NIH/NHLBI P01 Program Project: 1) demonstrate feasibility and participant acceptability of study design 2) demonstrate participant acceptability of measurement devices; 3) generate preliminary data to estimate outcome effect sizes.

In the course of WatchWell, the team of investigators will intervene on 3 behavioral mechanisms that are likely primary drivers of dSST CVD risk based on their prominent co-occurrence with rSST and individual contributions to CVD risk: blue light at night, nighttime food intake and prolonged evening sitting time. The investigators hypothesize that these 3 behavioral mechanisms impact CVD risk via downstream biological mechanisms including diurnal sleep/wake and body temperature rhythms, glucose metabolism, and autonomic balance (including heart rate variability, HRV). These biological mechanisms have not been assessed concurrently nor in the real-time, real-world context of rSST-related behaviors.

For this WorkWell pilot, the team of investigators will test 2 of the 3 behavioral mechanisms compared to the baseline control condition per participant using a 3-condition randomized controlled crossover design. [In the full trial to be resubmitted to the NIH, we will conduct a 4-condition crossover RCT, testing all 3 behavioral mechanisms compared to the baseline control condition per participant.] The investigators will recruit adults with overweight and at least 2 criteria of the metabolic syndrome (goal of N=18 completers, up to 30 enrollees total), who have elevated CVD risk. Impact. Recreational SST is a highly prevalent, modifiable risk factor for CVD. WorkWell will be the first to intervene on rSST-associated evening/nighttime blue light, food intake, and prolonged sitting in a real-world setting and to concurrently measure downstream CVD-related biological mechanisms. The WorkWell study design is informed by and will contribute to the translational application of circadian biology.

Aim 1. Assess the study feasibility and participant acceptability of delivering three behavioral strategies (avoiding dietary intake after 8p; blocking blue-light exposure after 8p; and breaking up prolonged sitting with standing after 5p) to reduce negative health exposures associated with rSST over two-week conditions in a randomized crossover study design.

Aim 2. Assess protocol compliance and participant acceptability of a suite of wearable sensors and home-based technologies during the feasibility trial.

Aim 3. Assess the preliminary efficacy and estimate effect size of the three behavioral strategies for improving postprandial glucose metabolism (primary focus on post-dinner meal, postprandial period), related 24-hr behaviors (sleep, other sedentary time, physical activity), heart rate variability, and circadian rhythms (sleep/wake activity rhythms, surface body temperature rhythms).

ELIGIBILITY:
Inclusion Criteria

* ≥26 years of age
* BMI ≥ 27 kg/m2*; ≥25 kg/m2, if Asian (full or multiple race)**
* Insufficiently active (per US National Guidelines for Physical Activity of 150 minutes of MVPA/Week)
* Reporting an average of ≥3 hours of recreational sedentary screen time (rSST) per day, that usually extends at least until 9:00pm.
* On a typical night, consumes calories (food and/or drink) after 8:00pm.
* Meet at least 2 criteria for metabolic syndrome

  * Central adiposity: waist circumference >40 inches (men); >35 inches (women)
  * Elevated blood pressure: SBP >130 mmHg and/or DBP >85 mmHg OR controlled with medication
  * Low high density lipoprotein (HDL) cholesterol: <40 mg/dL (men); <50 mg/dL (women)
  * Elevated triglycerides: >150 mg/dL OR controlled with medication
  * Elevated fasting glucose: ≥100 mg/dL OR controlled with medication

Exclusion Criteria

* Conditions related to sleep disruption, including lactation, pregnancy, mid-night care providers, sleep disorders, severe sleep apnea
* History of hypoglycemia
* Pacemaker
* Caffeine consumption in excess and/or after 5pm (excess equals >4 cups of coffee per day or equivalent)
* Involvement in other physical activity, diet, or weight loss programs/studies
* Weight change of 5% up or down in the last three months.
* Drug abuse
* THC use (smoking, edibles)
* Excessive alcohol use (for women, 8 or more drinks per week; for men, 15 or more drinks per week)
* Current smoker or user of any nicotine source - any amount or form (vapor/e-cig/tobacco/patch, gum, etc.)
* Medications that markedly impact glucose metabolism and sleep (insulin, corticosteroids, growth hormone, melatonin)
* Previous or current diagnosis of a clinical eating disorder (e.g., night eating syndrome, anorexia, bulimia, binge eating disorder); or self-report eating disorder behaviors
* Unstable or poorly controlled blood glucose (e.g., hypoglycemia, fasting glucose greater than 125 mg/dL)
* Chronic illness that may be associated with weight change (HIV/AIDS, active cancer, or uncontrolled thyroid disease)
* Shift work
* Recent or upcoming jetlag (travel 3 months prior and during study that is >1 time zone away from Arizona)
* Current practice of evening and nighttime blue light blocking.
* Poorly controlled hypertension (SBP ≥165 or DBP ≥100)
* Any condition or circumstance that would prevent compliance to the protocol
* Use non-android phone as their primary/personal phone

Min Age: 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment acceptability | 2 weeks
  Intervention acceptability will be assessed using the Treatment Evaluation Questionnaire (TEQ) to measure acceptability of the three experimental conditions following the completion of each condition. Scale Range: 0 to 4. Higher scores indicate greater acceptability.
Changes in Evening Sedentary Screen Time | 2 weeks
  Minutes per week of screen time after 5p as measured by WatchWell app and activPAL
Change in evening postprandial glycemic control (5pm - 5am) | 2 weeks
  Participants will be asked to wear the Dexcom G6 Pro continuous glucose monitor during baseline and experimental conditions. Glycemic control will be calculated by averaging all glucose readings from 5pm - 5am during each of the conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Sears, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided